CLINICAL TRIAL: NCT03170271
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo Controlled, Phase 3b Study to Evaluate the Safety and Efficacy of Benralizumab 30 mg sc in Patients With Severe Asthma Uncontrolled on Standard of Care Treatment
Brief Title: A Study of the Safety and Effectiveness of Benralizumab to Treat Patients With Severe Uncontrolled Asthma.
Acronym: ANDHI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3250C00045; 2017-001040-35 (EudraCT Number)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases; Additional relevant MeSH terms:; Asthma; Inflammation; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Pathologic Processes
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive; Inflammation; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Pathologic Processes | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Medi-563) (Experimental): Benralizumab (Medi563) Administered subcutaneously at Visit 4 (day 0), Visit 6 (day 28 +/- 3 days), Visit 7 (day 56 +/- 3 days) and Visit 9 (day 112 +/- 3 days) In the open label ANDHI IP sub study, all patients will receive benralizumab subcutaneously at Day 168 (Week 24), Day 196 (Week 28), Day 224 (Week 32), Day 280 (Week 40), Day 336 (Week 48), Day 392 (Week 56), Day 448 (Week 64), and Day 504 (Week 72).
  Interventions: Drug: Benralizumab (Medi-563)
- Placebo (Placebo Comparator): Administered subcutaneously at Visit 4 (day 0), Visit 6 (day 28 +/- 3 days), Visit 7 (day 56 +/- 3 days) and Visit 9 (day 112 +/- 3 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benralizumab (Medi-563) — 30mg Benralizumab administered as a subcutaneous injection at Visit 4 (day 0), Visit 6 (day 28 +/- 3 days), Visit 7 (day 56 +/- 3 days) and Visit 9 (day 112 +/- 3 days) In the open label ANDHI IP sub study, all patients will receive benralizumab subcutaneously at Day 168 (Week 24), Day 196 (Week 28), Day 224 (Week 32), Day 280 (Week 40), Day 336 (Week 48), Day 392 (Week 56), Day 448 (Week 64), and Day 504 (Week 72).
  Arms: Benralizumab (Medi-563)
Drug: Placebo — Placebo administered as a subcutaneous injection at Visit 4 (day 0), Visit 6 (day 28 +/- 3 days), Visit 7 (day 56 +/- 3 days) and Visit 9 (day 112 +/- 3 days)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of benralizumab on the rate of asthma exacerbations, patient reported quality of life and lung function during the 24-week treatment in patients with uncontrolled, severe asthma with an eosinophilic phenotype. A subset of patients will be assessed for their ongoing chronic rhinosinusitis with nasal polyps. The study design has been updated to include a 56-week open label ANDHI in Practice (ANDHI IP) sub study upon the completion of the 24-week double-blind period of the ANDHI study.

DETAILED DESCRIPTION:
This is a Phase IIIb, randomized, double-blind, placebo controlled, parallel group study designed to evaluate the efficacy and the safety of repeat dosing of benralizumab 30 mg subcutaneous (sc) versus placebo on top of standard of care asthma therapy in patients with severe uncontrolled asthma. Approximately 630 patients with peripheral blood eosinophil counts ≥150 cells/μL will be randomized 2:1 to receive benralizumab 30 mg sc or matched placebo for 24 weeks.

After enrolment, eligible patients will enter an up to 42-day screening/run-in period. Patients who meet eligibility criteria will be randomized 2:1 on Day 0 to receive either benralizumab or placebo every 56 days (every 8 weeks) through Week 16, with end of treatment (EOT) at Day 168 (Week 24). At the completion of the 24-week doubleblind period of the ANDHI study, eligible patients in benralizumab and placebo arm may enter a 56-week open label period (ANDHI in Practice [ANDHI IP] substudy), in which concomitant asthma therapies will be tapered as directed by the protocol in those patients who achieve and maintain asthma control (defined as ACQ6 score <1.5 and no clinically significant asthma exacerbations that required a burst of systemic corticosteroid or a hospitalization due to asthma between reduction visits) with add-on benralizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients aged 18 to 75 years inclusively at the time of Visit 1 with a history of physician-diagnosed asthma requiring treatment with medium-to-high dose Inhaled Corticosteroids (ICS) plus asthma controller, for at least 12 months prior to Visit 1.
2. Documented current treatment with high daily doses of ICS plus at least one other asthma controller for at least 3 months prior to Visit 1.
3. History of at least 2 asthma exacerbations while on ICS plus another asthma controller that required treatment with systemic corticosteroids (IM, IV, or oral) in the 12 months prior to Visit 1.
4. ACQ6 score ≥1.5 at Visit 1.
5. Screening pre-bronchodilator (pre-BD) FEV1 of <80% predicted at Visit 2.
6. Excessive variability in lung function by satisfying ≥ 1 of the following criteria:

   1. Airway reversibility (FEV1 ≥12%) using a short-acting bronchodilator demonstrated at Visit 2 or Visit 3.
   2. Airway reversibility to short-acting bronchodilator (FEV1 ≥12%) documented during the 12 months prior to enrolment Visit 1.
   3. Daily diurnal peak flow variability of >10% when averaged over 7 continuous days during the study run-in period
   4. An increase in FEV1 of ≥12% and 200 mL after a therapeutic trial of systemic corticosteroid (eg, OCS), given outside of an asthma exacerbation, documented in the 12 months prior enrolment Visit 1.
   5. Airway hyper-responsiveness (methacholine: PC20 of <8 mg/mL, histamine: PD20 of <7.8 μmol, mannitol: decrease in FEV1 as per the labelled product instructions) documented in the 24 months prior to randomization Visit 4.
7. Peripheral blood eosinophil count either:

   * 300 cells/μL assessed by central laboratory at either Visit 1 or Visit 2

OR

≥150 to <300 cells/μL assessed by central laboratory at either Visit 1 or Visit 2, IF ≥1 of the following 5 clinical criteria (a to e) is met:

1. Using maintenance OCS (daily or every other day OCS requirement in order to maintain asthma control; maximum total daily dose 20 mg prednisone or equivalent) at screening
2. History of nasal polyposis
3. Age of asthma onset ≥18 years
4. Three or more documented exacerbations requiring systemic corticosteroid treatment during the 12 months prior to screening
5. Pre-bronchodilator forced vital capacity <65% of predicted, as assessed at Visit 2 (note that screening pre-BD FEV1 Inclusion Criterion #6 must still be satisfied)

For inclusion in the open label ANDHI IP sub study patients should meet the following criteria:

1. Patients study must have completed ANDHI EOT Visit 11.
2. Written informed consent must also be obtained prior to any study related procedures being performed in the open label ANDHI IP sub study.
3. Patients who have received any approved or investigational targeted biologic for the treatment of asthma (e.g. commercial mepolizumab, reslizumab, benralizumab) may be included if the last dose is ≥ 2 months of Visit 13.

Exclusion Criteria:

1. Clinically important pulmonary disease other than asthma
2. Acute upper or lower respiratory infections within 30 days prior to the date informed consent.
3. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy.
4. History of alcohol or drug abuse within 12 months prior to the date informed consent is obtained.
5. A history of known immunodeficiency disorder.
6. Current smokers or former smokers with a smoking history of ≥10 pack years.
7. Previously received benralizumab (MEDI-563).
8. Receipt of any investigational medication as part of a research study within approximately 5 half-lives prior to randomization.
9. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
10. Receipt of live attenuated vaccines 30 days prior to the date of randomization; other types of vaccines are allowed.
11. Concurrent enrolment in another interventional or post-authorization safety study

Exclusion criteria for the open label ANDHI IP sub study:

Patients should not enter the open label ANDHI IP sub study if any of the following exclusion criteria are fulfilled. Each exclusion criterion should be reviewed in all potential participants, including those who transition directly from the double-blind period and those with a delay between completing the EOT Visit 11 and the first open label visit (Visit 13).

1. Patients who participated in the double-blind period but failed to complete the ANDHI EOT Visit 11. Patients who completed the ANDHI FU Visit 12 are not excluded from participation in the ANDHI IP sub study.
2. Unable to commit to the monthly visits as required by the protocol, or unable to commit to undergoing protocol guided reductions in asthma therapy, as directed by the Investigator.
3. Patients who experienced a severe or serious treatment-related AE during the double-blind period and, and those whom Investigator judges it is not in the patient's best interest to extend possible treatment with benralizumab.
4. Approved or off-label use of systemic immunosuppressive medications within 3 months prior to the first open label visit (Visit 13). These include but are not limited to small molecules such as methotrexate, cyclosporine, azathioprine, and immunosuppressive/immunomodulating biologics such as tumour necrosis factor (TNF) blockers. Regular use of systemic OCS is also excluded except for the indication of asthma.
5. Receipt of live attenuated vaccines 30 days prior to the first visit in the open label ANDHI IP sub study (Visit 13); other types of vaccines are allowed.
6. Planned surgical procedures during the conduct of the study.
7. Positive urine pregnancy test at Visit 13, or currently breastfeeding or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Goodman, MD, Principal Investigator — Aero Allergy Research Lab of Savannah; Vinay Sikand, MD, Principal Investigator — Sikand Institute of Pulmonary Research; Willaim Cherry, MD, Principal Investigator — Riverside Medical Center
Locations (199):
- United States (90):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Encinitas, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, South Bend, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Lakeside Park, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Chevy Chase, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Highland Park, New Jersey
  - Research Site, Marlton, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, Piscataway, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Grove City, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Clackamas, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Franklin, Tennessee
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Galveston, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Provo, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, North Chesterfield, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Everett, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, West Allis, Wisconsin
- Austria (2):
  - Research Site, Feldbach
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Liège
  - Research Site, Montigny-le-Tilleul
  - Research Site, Namur
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (3):
  - Research Site, Aarhus N
  - Research Site, Odense C
  - Research Site, Vejle
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Turku
- France (21):
  - Research Site, Bayonne
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, La Roche-sur-Yon
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Marburg
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Rheine
  - Research Site, Rüdersdorf
  - Research Site, Wangen
- Italy (20):
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cona
  - Research Site, Foggia
  - Research Site, Garbagnate Milanese
  - Research Site, Legnago
  - Research Site, Matera
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Piacenza
  - Research Site, Pietra Ligure
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Verona
- Netherlands (7):
  - Research Site, Amersfoort
  - Research Site, Deventer
  - Research Site, Enschede
  - Research Site, Harderwijk
  - Research Site, Helmond
  - Research Site, Nijmegen
  - Research Site, Zwolle
- Norway (2):
  - Research Site, Bergen
  - Research Site, Lørenskog
- Spain (15):
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Jerez de la Frontera
  - Research Site, Laredo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Taco
  - Research Site, Valdemoro
- Sweden (3):
  - Research Site, Lund
  - Research Site, Östersund
  - Research Site, Stockholm
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Louis R, Harrison TW, Chanez P, Menzella F, Philteos G, Cosio BG, Lugogo NL, de Luiz G, Burden A, Adlington T, Keeling N, Kwiatek J, Garcia Gil E; ANDHI Study Investigators. Severe Asthma Standard-of-Care Background Medication Reduction With Benralizumab: ANDHI in Practice Substudy. J Allergy Clin Immunol Pract. 2023 Jun;11(6):1759-1770.e7. doi: 10.1016/j.jaip.2023.03.009. Epub 2023 Mar 21. PMID 36948488
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- [Derived] Harrison TW, Chanez P, Menzella F, Canonica GW, Louis R, Cosio BG, Lugogo NL, Mohan A, Burden A, McDermott L, Garcia Gil E, Zangrilli JG; ANDHI study investigators. Onset of effect and impact on health-related quality of life, exacerbation rate, lung function, and nasal polyposis symptoms for patients with severe eosinophilic asthma treated with benralizumab (ANDHI): a randomised, controlled, phase 3b trial. Lancet Respir Med. 2021 Mar;9(3):260-274. doi: 10.1016/S2213-2600(20)30414-8. Epub 2020 Dec 22. PMID 33357499
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00045&attachmentIdentifier=9ee3eb1e-53ba-4b2b-8800-1dd44269f23a&fileName=D3250C00045_CSP_v4.0_Final_22SEP20_Redacted_PDFA.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00045&attachmentIdentifier=b0e85ad9-7be7-42a2-ace7-8aa882732f3a&fileName=D3250C00045_SAP_ed3.0_Final_22SEP20_Redacted_PDFA.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00045&attachmentIdentifier=b445a28c-2828-42a1-813d-19218e2ca383&fileName=D3250C00045-CSR_synopsis-ANDHI_Main_Final_Redacted_19Oct21_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with severe uncontrolled asthma and peripheral blood eosinophil counts of ≥150 cells/microliter (μL) (with major subgroups of 150-300 cells/μL plus clinical features and ≥300 cells/μL) were recruited to 221 centers in 14 countries. Patients were randomized in a 2:1 ratio to receive benralizumab or matched placebo for 24 weeks. Results are reported for the double-blind period of the study (data cut-off: 12 Sep 2019).
Pre-assignment Details: Severe eosinophilic patients were to have had ≥ 2 asthma exacerbations while on maintenance inhaled corticosteroids (ICS) plus another asthma controller that required treatment with systemic corticosteroids in the 12 months prior to enrolment. Patients continued to receive their standard of care asthma therapy throughout the study period.
Groups:
- Benralizumab: Patients received benralizumab 30 milligrams (mg) administered subcutaneously (sc) in an accessorized pre-filled syringe at Week 0 (initial dose), Week 4 (loading dose), Week 8 and Week 16. An End of Treatment (EOT) visit was performed at Week 24.
- Placebo: Patients received matching placebo solution administered sc in an accessorized pre-filled syringe at Week 0 (initial dose), Week 4 (loading dose), Week 8 and Week 16. An EOT visit was performed at Week 24.
Period: Overall Study
Arm/Group | Benralizumab | Placebo
Started (Randomized) | 431 | 229
Received Treatment | 427 | 229
Completed (Completed double-blind period of study) | 398 | 218
Not Completed | 33 | 11
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol-specified withdrawal criterion | 2 | 1
Not completed — Withdrawal by Subject | 17 | 5
Not completed — Other | 2 | 2
Not completed — Randomized in error | 4 | 0

BASELINE CHARACTERISTICS:
Population: All patients in the full analysis set (FAS) who received any investigational product (IP) were included in the baseline analysis.
Groups:
- Benralizumab: Patients received benralizumab 30 mg administered sc in an accessorized pre-filled syringe at Week 0 (initial dose), Week 4 (loading dose), Week 8 and Week 16. An EOT visit was performed at Week 24.
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo | Total
Number analyzed (Participants) | 427 | 229 | 656
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (12.69) | 53.3 (12.52) | 52.8 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 136 | 399
  Male | 164 | 93 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 25 | 74
  Not Hispanic or Latino | 318 | 172 | 490
  Unknown or Not Reported | 60 | 32 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 314 | 168 | 482
  Black or African American | 35 | 18 | 53
  Asian | 11 | 7 | 18
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Other | 5 | 2 | 7
  Missing | 62 | 33 | 95
Screening eosinophil count group (cells/µL) [Count of Participants; unit: Participants]
  ≥ 150 - < 300 | 129 | 63 | 192
  ≥ 300 | 297 | 165 | 462
  Missing | 1 | 1 | 2
Baseline eosinophil count group (cells/μL) [Count of Participants; unit: Participants]
  < 300 | 146 | 74 | 220
  ≥ 300 - < 450 | 105 | 56 | 161
  ≥ 450 | 176 | 99 | 275

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Asthma Exacerbations Over the Treatment Period (up to Week 24)
Description: An asthma exacerbation was defined as a worsening of asthma that led to any of the following:
  * Use of systemic corticosteroids (or temporary increase in stable oral corticosteroids [OCS] background dose) for at least 3 days; a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of systemic corticosteroids.
  * An emergency room/urgent care visit (defined as evaluation and treatment for < 24 hours in an emergency department or urgent care center) due to asthma that required systemic corticosteroids (as per above).
  * An inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥ 24 hours) due to asthma.
  Annual exacerbation rate = 365.25*total number of exacerbations / total duration of follow-up within the treatment group. Annual asthma exacerbation rates over the 24-week period were estimated using a negative binomial model.
Time Frame: Baseline (Week 0) up to Week 24
Population: The FAS included all randomized patients who received at least 1 dose of IP, irrespective of their protocol adherence and continued participation in the study.
Measure: Number (95% Confidence Interval); unit: Events/year
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 427 | 229
Events/year | 0.94 [0.79 to 1.12] | 1.86 [1.54 to 2.24]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Comparison of annual exacerbation rates for benralizumab vs placebo (rate ratio). Treatment group, region, number of exacerbations in previous year and maintenance OCS use at baseline were included in the negative binomial model as covariates. The log of each patient's corresponding follow-up time was used as an offset variable in the model to adjust for patients having different follow-up times during which events occurred; Test type: Superiority — The null hypothesis was that the exacerbation rate of benralizumab was equal to the exacerbation rate of placebo; p < 0.0001, Negative binomial; Rate ratio = 0.51, 95% CI 2-sided [0.39 to 0.65]

2. Secondary Outcome: Change From Baseline in Saint George Respiratory Questionnaire (SGRQ) Total Score to the EOT (Week 24)
Description: The SGRQ is a 50-item patient-reported outcome instrument which measures the health status of patients with airway obstruction diseases. The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The SGRQ total score indicates the impact of disease on overall health status and is expressed as a percentage of overall impairment (scores range from 0 to100, with 100 representing worst possible health status and 0 indicating the best possible health status). The least squares (LS) mean change from baseline in SGRQ total score at Week 24 is presented.
Time Frame: Baseline (Week 0) and Week 24
Population: The FAS included all randomized patients who received at least 1 dose of IP, irrespective of their protocol adherence and continued participation in the study. Only patients with data available at the timepoints of testing were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 364 | 204
Scores on a scale | -23.06 (1.00) | -14.94 (1.34)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in SGRQ total score at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a mixed-effect model for repeated measures (MMRM) analysis; Test type: Superiority; p < 0.0001, Repeated measures analysis; LS Mean difference = -8.11, 95% CI 2-sided [-11.41 to -4.82] — Model: Change from baseline in SGRQ total score = Treatment + baseline SGRQ total score + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit

3. Secondary Outcome: Change From Baseline in Pre-Bronchodilator (BD) Forced Expiratory Volume in First Second (FEV1) to the EOT (Week 24)
Description: Lung function was assessed by FEV1 which was measured by spirometry. Spirometry was performed by the Investigator or authorized delegate according to American Thoracic Society/European Respiratory Society guidelines. The LS mean change from baseline in pre-BD FEV1 at Week 24 is presented.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 393 | 213
Liters (L) | 0.30 (0.02) | 0.14 (0.03)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in pre-BD FEV1 at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p < 0.0001, Repeated measures analysis; LS Mean difference = 0.16, 95% CI 2-sided [0.09 to 0.23] — Model: Change from baseline in pre-BD FEV1 = Treatment + baseline pre-BD FEV1 + region + number of exacerbations in previous year + maintenance OCS use at baseline + gender + age + visit + treatment by visit

4. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 6 (ACQ-6) Score to the EOT (Week 24)
Description: The ACQ-6 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath and wheezing) and short-acting β-2 receptor agonist use. Patients were asked to recall the status of their asthma during the previous week and respond to the questions of the ACQ-6 on a 7-point scale. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is computed as the mean of the responses from all the items in the questionnaire. Mean scores of ≤0.75 indicated well-controlled asthma, scores between 0.75 and <1.5 indicated partly-controlled asthma, and a score ≥1.5 indicated not well-controlled asthma. The LS mean change from baseline in ACQ-6 score at Week 24 is presented.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 393 | 216
Scores on a scale | -1.47 (0.06) | -1.01 (0.08)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in ACQ-6 score at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p < 0.0001, Repeated measures analysis; LS Mean difference = -0.46, 95% CI 2-sided [-0.65 to -0.27] — Model: Change from baseline in ACQ-6 score = Treatment + baseline ACQ-6 score + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit

5. Secondary Outcome: Time to First Asthma Exacerbation (up to Week 24)
Description: Time to first asthma exacerbation was derived as follows:
  Start date of first asthma exacerbation - Date of randomization + 1. The time to first asthma exacerbation for patients who did not experience an asthma exacerbation during the treatment period was censored at the EOT visit (Week 24) for patients who completed the study. Patients who withdrew from the study or were lost to follow-up before the EOT visit were censored at the last visit date after which an exacerbation could not be assessed. The median time to first asthma exacerbation was not calculated, so the number of patients who experienced an asthma exacerbation is presented for the measured values.
Time Frame: Baseline (Week 0) up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 427 | 229
Participants | 123 | 107
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Comparison of time to first asthma exacerbation for benralizumab vs placebo. Treatment group, region, number of exacerbations in previous year and maintenance OCS use at baseline were included in the Cox proportional hazard model as covariates; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.40 to 0.67] — A hazard ratio < 1 favours benralizumab to be associated with a longer time from randomization to the first exacerbation than placebo

6. Secondary Outcome: Change From Run-in Baseline Home Peak Expiratory Flow (PEF) (Morning and Evening) to the EOT (Week 24)
Description: Home PEF testing was performed by the patient each morning after awakening and before taking their morning asthma medications, and each evening using a peak flow meter. Measurements were taken at approximately the same time each day and recorded in the Asthma Daily Diary. The maximum of the 3 measurements performed every morning and evening were used in the calculation of the weekly means. A weekly mean was calculated as the sum of all non-missing daily measures over the 7 sequential days divided by the number of non-missing daily measures. If more than 3 daily measures (> 50%) within a period were missing, then the weekly mean for that period was set to 'missing'. Change from run-in baseline in weekly means for morning PEF and evening PEF are presented. Baseline was the average for data collected over the last 7 days of the run-in period prior to randomization.
Time Frame: Run-in baseline (from Day -28 to Day 0) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: L/minute
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 427 | 229
L/minute
  Morning: number analyzed (Participants) | 276 | 142
  Morning | 27.17 (3.98) | 7.06 (5.49)
  Evening: number analyzed (Participants) | 256 | 144
  Evening | 16.47 (4.04) | -6.61 (5.54)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from run-in baseline in morning PEF at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0031, Repeated measures analysis; LS Mean difference = 20.11, 95% CI 2-sided [6.79 to 33.44] — Model: Change from baseline in PEF = Treatment + baseline PEF + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Change from run-in baseline in evening PEF at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0008, Repeated measures analysis; LS Mean Difference = 23.09, 95% CI 2-sided [9.62 to 36.55] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in Short Form 36-item Health Survey, Version 2 (SF-36v2) to the EOT (Week 24)
Description: The SF-36v2 is a 36-item survey of functional health and well-being, with a 1 week recall period. The 8-domain profile consists of the following subscales: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The physical and mental health component summary scores are computed from subscale scores to give a broader metric of physical and mental health-related quality of life. Each domain score, as well as the physical and mental component scores, were scored on a scale from 0-100 (worst health possible to best health possible); higher scores indicate better health status. Norm-based scoring was used to calculate the 8 SF-36v2 subscales and the 2 component scores. The LS mean change from baseline in each of the SF-36 subscale and component summary scores at Week 24 are presented.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 287 | 169
Scores on a scale
  Physical functioning | 17.76 (1.21) | 12.42 (1.59)
  Role limitations due to physical health | 17.62 (1.34) | 10.82 (1.76)
  Bodily pain | 6.44 (1.37) | 3.37 (1.79)
  General health perceptions | 12.92 (1.01) | 7.29 (1.34)
  Vitality | 12.04 (1.10) | 6.53 (1.44)
  Social functioning | 12.44 (1.34) | 9.32 (1.75)
  Role limitations due to emotional problems | 8.23 (1.18) | 5.79 (1.55)
  Mental health | 5.57 (0.90) | 3.89 (1.18)
  Physical health component summary score | 6.09 (0.46) | 3.77 (0.60)
  Mental health component summary score | 2.87 (0.48) | 1.99 (0.64)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for physical functioning at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0077, Repeated measures analysis; LS Mean difference = 5.35, 95% CI 2-sided [1.42 to 9.28] — Model: Change from baseline in SF-36v2 score = Treatment + baseline SF-36v2 score + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for role limitations due to physical health at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0022, Repeated measures analysis; LS Mean Difference = 6.80, 95% CI 2-sided [2.45 to 11.14] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for bodily pain at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.1741, Repeated measures analysis; LS Mean Difference = 3.07, 95% CI 2-sided [-1.36 to 7.50] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for general health perceptions at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0009, Repeated measures analysis; LS Mean Difference = 5.62, 95% CI 2-sided [2.32 to 8.92] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for vitality at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0025, Repeated measures analysis; LS Mean Difference = 5.51, 95% CI 2-sided [1.95 to 9.08] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for social functioning at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.1583, Repeated measures analysis; LS Mean Difference = 3.12, 95% CI 2-sided [-1.22 to 7.46] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for role limitations due to emotional problems at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.2103, Repeated measures analysis; LS Mean Difference = 2.44, 95% CI 2-sided [-1.38 to 6.27] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 8: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 subscale score for mental health at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.2581, Repeated measures analysis; LS Mean Difference = 1.68, 95% CI 2-sided [-1.23 to 4.59] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 physical health component summary score at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0022, Repeated measures analysis; LS Mean Difference = 2.32, 95% CI 2-sided [0.84 to 3.81] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 10: Comparison: Benralizumab vs Placebo; Change from baseline in SF-36v2 mental health component summary score at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.2751, Repeated measures analysis; LS Mean Difference = 0.87, 95% CI 2-sided [-0.70 to 2.44] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Patient Global Impression of Severity (PGI-S): Responder Status at the EOT (Week 24)
Description: The PGI-S is a single question asking the patient to rate the overall severity of their symptoms using a 6-point categorical response scale from 0 to 5 where 0=no symptoms and 5=very severe symptoms. Higher scores indicate a worse outcome. Improvement was defined as a PGI-S at EOT (Week 24) better than PGI-S at baseline. Important improvement was defined as PGI-S at baseline = moderate symptoms or severe symptoms or very severe symptoms shifting to PGI-S at EOT = no symptoms or very mild symptoms or mild symptoms. Patients with missing data at the EOT visit who did not complete the study were considered non-responders. For patients who completed the study with missing data at EOT (Week 24), their last evaluable post-baseline score was used to define responder status. The percentage of patients for each of the indicated PGI-S responder categories are presented.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 345 | 187
Percentage of patients
  Improvement | 61.7 | 53.5
  Important improvement | 45.5 | 38.0
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a responder classified as type 'Improvement' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p = 0.0233, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.06 to 2.25] — Model: ln (1/(1-p)) = Treatment + baseline score + region + number of exacerbations in previous year + maintenance OCS use at baseline, where p is the proportion of patients being a responder
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a responder classified as type 'Important Improvement' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p = 0.0401, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.02 to 2.16] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Clinician Global Impression of Change (CGI-C) and Patient Global Impression of Change (PGI-C): Responder Status at the EOT (Week 24)
Description: The Investigator (clinician) and the patient were asked separately to rate the degree of change in the overall asthma status compared to the start of treatment, i.e. baseline randomization visit. A 7-point rating scale was used for the CGI-C (rated by Investigator) and PGI-C (rated by patient) where: 1=Very Much Improved; 2=Much Improved; 3=Minimally Improved; 4=No Changes; 5=Minimally Worse; 6=Much Worse, and 7=Very Much Worse. Higher scores indicate a worse outcome. Responder category definitions: Much improved = (Much improved, Very much improved); Very much improved = (Very much improved). Patients with missing data at the EOT visit who did not complete the study were considered non-responders. For patients who completed the study with missing data at EOT (Week 24), their last evaluable post-baseline score was used to define responder status. The percentage of patients for each of the indicated CGI-C and PGI-C responder categories are presented.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 427 | 229
Percentage of patients
  CGI-C: Much improved: number analyzed (Participants) | 420 | 227
  CGI-C: Much improved | 52.9 | 35.2
  CGI-C: Very much improved: number analyzed (Participants) | 420 | 227
  CGI-C: Very much improved | 15.0 | 4.8
  PGI-C: Much improved: number analyzed (Participants) | 424 | 228
  PGI-C: Much improved | 55.9 | 38.2
  PGI-C: Very much improved: number analyzed (Participants) | 424 | 228
  PGI-C: Very much improved | 37.7 | 16.7
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a CGI-C responder classified as type 'Much improved' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.47 to 2.86] — Model: ln (1/(1-p)) = Treatment + region + number of exacerbations in previous year + maintenance OCS use at baseline, where p is the proportion of patients being a responder
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a CGI-C responder classified as type 'Very much improved' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.77 to 6.70] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a PGI-C responder classified as type 'Much improved' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.48 to 2.87] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Benralizumab vs Placebo; Estimate of the log odds of being a PGI-C responder classified as type 'Very much improved' at Week 24 in the benralizumab group compared to the placebo group using a logistic regression; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.02, 95% CI 2-sided [2.02 to 4.51] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Predominant Symptom and Impairment Assessment (PSIA) Severity Score for Average of Top 3 Ranked Symptoms/Impairments and for Top Ranked Symptom/Impairment at the EOT (Week 24)
Description: For part 1 of the PSIA only administered at baseline, patients reviewed 8 concepts (including cardinal asthma symptoms, activities, awakenings, triggers) and selected those which were typically bothersome. Based on part 1 selections, part 2 of the PSIA produced a rank ordered list of bothersome concepts individualized per the patient for subsequent evaluation. For part 3 of the PSIA assessed at baseline and during the study, patients recorded the severity of each selected symptom or impairment using an 11-point numeric rating scale where: 0=Did not experience and 10=Worst I can imagine. Higher scores indicate a worse outcome. The LS mean change from baseline in PSIA severity score for the indicated categories at Week 24 are presented. A negative change from baseline indicates an improvement in symptoms. Note: Average PSIA was calculated only where all of top 3 ranked symptoms/impairments were available, otherwise average was set to missing.
Time Frame: Baseline (Week 0) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 319 | 180
Scores on a scale
  Average of top 3 ranked: number analyzed (Participants) | 302 | 172
  Average of top 3 ranked | -2.97 (0.14) | -1.82 (0.19)
  Top ranked | -3.02 (0.15) | -1.87 (0.20)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in PSIA severity score for the average of top 3 ranked symptoms/impairments at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p < 0.0001, Repeated measures analysis; LS Mean difference = -1.15, 95% CI 2-sided [-1.62 to -0.68] — Model: Change from baseline in average PSIA score (top 3 ranked) =Treatment + baseline average PSIA score (top 3 ranked) + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Change from baseline in PSIA severity score of top ranked symptom/impairment at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p < 0.0001, Repeated measures analysis; LS Mean difference = -1.15, 95% CI 2-sided [-1.64 to -0.66] — Model: Change from baseline in PSIA score (top ranked) =Treatment + baseline PSIA score (top ranked) + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit

11. Secondary Outcome: Change From Baseline in the Sino-Nasal Outcome Test Item 22 (SNOT-22) Total Score to the EOT (Week 24)
Description: The 22-item SNOT 22 questionnaire was used to assess the rhinosinusitis health status and quality of life of patients with baseline chronic rhinosinusitis with nasal polyposis. The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110. Higher scores indicate poorer outcomes. The LS mean changes from baseline in SNOT-22 total score in patients in the chronic rhinosinusitis with nasal polyposis sub-study analysis set at Week 24 are presented.
Time Frame: Baseline (Week 0) and Week 24
Population: The chronic rhinosinusitis with nasal polyposis sub-study analysis set was defined as the subset of patients with doctor-diagnosed chronic rhinosinusitis and nasal polyposis included in their medical history who had signed the informed consent to participate in the sub-study and who had received at least 1 dose of IP.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 92 | 50
Scores on a scale | -19.02 (2.27) | -10.11 (3.04)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Change from baseline in SNOT-22 total score at Week 24 was compared between the benralizumab group and placebo group using a restricted maximum likelihood based on a MMRM analysis; Test type: Superiority; p = 0.0204, Repeated measures analysis; LS Mean difference = -8.91, 95% CI 2-sided [-16.42 to -1.40] — Model: Change from baseline in SNOT-22 total score = Treatment + baseline SNOT-22 total score + region + number of exacerbations in previous year + maintenance OCS use at baseline + visit + treatment by visit

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data is reported for the on-treatment period + follow-up (up to a maximum of 24 weeks). Assessed until 12 Sep 2019 analysis cut-off date.
Description: AE definition for on-treatment period: onset date ≥ first dose of IP and ≤ scheduled EOT visit, or IP discontinuation (IPD) visit for patients prematurely discontinuing IP. If both EOT and IPD visits were missing, upper limit of the on-treatment period was defined as day of last dose of IP + 56 days. If upper limit was after end of the on-study period, upper limit was set to end of on-study period.
Arm/Group | Benralizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/427 | 0/229
Serious Adverse Events (participants affected / at risk) | 23/427 | 25/229
Other Adverse Events (participants affected / at risk) | 136/427 | 78/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=427) | Placebo (N=229)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=427) | Placebo (N=229)
Pyrexia (General disorders) | 26 (29) | 5 (8)
Bronchitis (Infections and infestations) | 22 (23) | 18 (22)
Nasopharyngitis (Infections and infestations) | 30 (36) | 17 (23)
Sinusitis (Infections and infestations) | 28 (32) | 12 (17)
Upper respiratory tract infection (Infections and infestations) | 17 (19) | 12 (13)
Headache (Nervous system disorders) | 37 (50) | 7 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 13 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 13 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03170271/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT03170271/SAP_002.pdf